CLINICAL TRIAL: NCT03922087
Title: Huizhou Mother-infant Cohort
Brief Title: No-worry Baby Project
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Huizhou No.1 Maternal and Child Care Service Cencer (Unknown)
Responsible Party: Principal Investigator, LIU ZHAOMIN, Professor in Department of Nutrition and Food Hygiene, Sun Yat-sen University
Other Study IDs: HZT2018
Record Dates: First submitted 2019-04-13; First posted 2019-04-19 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Gestational Hypertension; Thyroid Disease Pregnancy; Obesity; Anemia in Pregnancy; Complications, Pregnancy; Depression; Obstetric Labor Complications; Asthma; Allergic Disorder; Immune System Diseases; Neurodevelopmental Disorders; Reproductive Disorder
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Obesity; Pregnancy Complications; Depression; Obstetric Labor Complications; Asthma; Hypersensitivity; Immune System Diseases; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During pregnancy: maternal vein blood at mid- and last trimester, spot and 12-hr urine and feces at mid-trimester; At delivery: umbilical cord blood, placenta , umbilical cord, mother's milk. Postnatal: mother's vein blood During infancy: meconium. During childhood: Mother's milk and baby's feces.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: The pregnancy women without any diseases.
  Interventions: Other: No intervention
- Disease Group: The pregnancy women with cardio-metabolic and endocrinic disorders such as gestational diabetes, obesity, hypertension, thyroid diseases, anemia and other cardio-metabolic diseases.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The Huizhou mother-infant cohort was set up to investigate the effect of dietary factors and environmental exposures during pregnancy on health consequences of mothers and offsprings in Huizhou, China.

DETAILED DESCRIPTION:
Huizhou mother-infant cohort (No-worry Baby Project) is a scientific research/public health project jointly initiated by Huizhou First Maternity and Child Healthcare Hospital and School of Public Health, Sun Yat-sen University. The project plans to recruit 10,000 participants since early pregnancy and follow up for three years after birth in the first stage. Biological samples, data from questionnaires survey and clinical information will be collected for both mothers and infants. The study is aimed to investigate the effects of dietary factors and environmental exposures during pregnancy on infants' health as well as the prognosis of diseased mothers. The study will have essentially both clinical and public health implications to find effective strategies for prevention and management of a range of chronic disorders (above mentioned) during pregnancy and exploration of the possible impacts on offspring health. The cohort will provide scientific basic for improvement of mother and infant's health.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who have plan to delivery and participate in child care in Huizhou hospital;
* Pregnant women who have resided in Huizhou for at least 3 years;
* Pregnant women who are consent for specimens and data collection and follow-ups for both mother and infant.

Exclusion Criteria:

* Pregnant women who are with gestational age more than 24 weeks ;
* Pregnant women who refuse to participate or be unwilling to sign informed consent;
* Pregnant women who are mentally incapacitated and need guardians.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eligible pregnant women will be recruited from Huizhou First Maternal and Child Care Service Center.
Sampling Method: Probability Sample
Enrollment: 5216 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Number of adverse birth outcomes. | At delivery.
  Including dystocia,stillbirth, fetal macrosomia and child with birth defect.
Children weight changes. | At age of 1 month, 3 months, 6months, 1 year, and 3 year.
  Weight is measured in kilograms.
Children height changes. | At age of 1 month, 3 months, 6months, 1 year, and 3 year.
  Height is measured in meters.
Number of participant with gestational complications. | At delivery.
  Including gestational hypertension and preeclampsia, and gestational diabetes mellitus.

SECONDARY OUTCOMES:
Maternal weight changes(kg). | At 20 weeks of gestation, 28 weeks of gestation, the time before labor and 30 days after delivery.
  Assess using electronic weighing machine and body composition analyzer.
Number of participant with postnatal depression. | At 30 days after delivery.
  Assess using Edinburgh Postnatal Depression Scale (EPDS). The total score of scale is 30 ,and higher score indicates worse status.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaomin Liu, Doctor, Principal Investigator — School of Public Health of Sun Yat-sen University
Locations (1):
- School of Public Health of Sun Yat-sen University (North Campus), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu ZM, Long HH, Li D, Fang AP, Chen CG, Wang C, Li MM, Wu Y, Zhang SJ, Pan WJ. Maternal Serum Iodine Concentrations in Early Pregnancy Exhibited Well Diagnostic Ability for Thyroid Dysfunction, Inverse Associations with Gestational Weight Gain, and Birth Size: Longitudinal Analyses Based on Huizhou Mother-Infant Cohort. Biol Trace Elem Res. 2025 Jul;203(7):3618-3629. doi: 10.1007/s12011-024-04443-7. Epub 2024 Nov 29. PMID 39609361
- [Derived] Zhang D, Zhang S, Li G, Lai Y, Hao YT, Chen WQ, Wu Y, Chen C, Pan W, Liu ZM. A clinical model and nomogram for early prediction of gestational diabetes based on common maternal demographics and routine clinical parameters. J Obstet Gynaecol Res. 2022 Nov;48(11):2738-2747. doi: 10.1111/jog.15380. Epub 2022 Jul 31. PMID 35909297